CLINICAL TRIAL: NCT01336530
Title: Clinical Trial to Assess the Efficacy of Fixed Combination Product Tepilta® in the Treatment of Radiation-induced Oesophagitis Compared to Its Active Ingredients Oxetacaine and Antacids, and to Placebo
Brief Title: Tepilta® Versus Oxetacaine, Antacids and Placebo
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study stopped prematurely due to and administrative reasons, not based on grounds of safety.
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: Trium Analysis Online GmbH (Industry); ICON plc (Industry); Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: X-03030-3277; 2009-014441-93 (EudraCT Number)
Record Dates: First submitted 2011-04-01; First posted 2011-04-18 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2017-02

CONDITIONS: Radiation-induced Oesophagitis
Keywords: Oesophageal pain; Radiotherapy; Combined radio-chemotherapy; Oesophageal symptoms
MeSH Terms: interventions — oxethazaine; Aluminum; Magnesium Hydroxide; Magnesium; Aluminum Hydroxide; Antacids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tepilta® (Experimental)
  Interventions: Drug: oxetacaine, aluminium and magnesium hydroxide
- Oxetacaine (Active Comparator)
  Interventions: Drug: oxetacaine
- Antacids (Active Comparator)
  Interventions: Drug: magnesium and aluminium hydroxide
- Placebo (Placebo Comparator)
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: oxetacaine, aluminium and magnesium hydroxide — 20mg/10ml oxetacaine, 196mg/10ml magnesium hydroxide, 582mg/10ml aluminium hydroxide. Suspension for oral intake 3-6 times per day for a maximum of 11 weeks.
  Other Names: Tepilta®
  Arms: Tepilta®
Drug: oxetacaine — 20mg/10ml oxetacaine. Suspension for oral intake 3-6 times per day for a maximum of 11 weeks.
  Arms: Oxetacaine
Drug: magnesium and aluminium hydroxide — 196mg/10ml magnesium hydroxide, 582mg/10ml aluminium hydroxide. Suspension for oral intake 3-6 times per day for a maximum of 11 weeks.
  Other Names: Antacids
  Arms: Antacids
Other: Vehicle — Placebo suspension for oral intake 3-6 times per day for a maximum of 11 weeks.
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled, therapeutic confirmatory multicentre trial with 4 parallel treatment groups. The design is adaptive group-sequential with two interim analyses, possible sample size re-estimation after the first or second interim analysis and drop-the-loser approach. The study design was primarily chosen to show superior efficacy of Tepilta® compared to the single components and to placebo. Evaluation of safety is a secondary objective.

DETAILED DESCRIPTION:
Tepilta® Suspension is indicated for treatment of pain in the upper digestive system induced by radiation therapy, in particular for radiation-induced oesophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years.
2. Score = 0 on NRS for oesophageal pain.
3. Radiotherapy (RT) or combined radio-chemotherapy (RCT) of a solid tumour in head/neck/thorax region. A minimum length of 5 cm of the oesophagus must be included in high-dose radiation field.
4. Duration of RT 5 to 8 weeks.
5. Single radiation dosage of fractionated RT 1.8 to 2.0 Gy/day, of intensity-modulated RT (IMRT) 1.5 to 2.3 Gy/day, each for 5 days a week (single frequency deviations are allowed presuming that intended duration of RT remains 5 to 8 weeks).
6. First radiation in the intended radiation area.
7. Written informed consent.

   Randomisation criteria:
8. Appearance of oesophageal pain as follows: Score ≥ 2 on Numeric Rating Scale (NRS) for pain during main daily meals is reached at least once.
9. At least 20 Gy of the dose of radiation therapy in oesophageal area remaining.
10. Oesophageal symptoms of grade ≤ 2a according to the adapted Common Terminology Criteria for Adverse Events CTCAE.

Exclusion Criteria:

1. History of allergic reaction to the study medication or its excipients (i.e. aluminium or magnesium hydroxide, oxetacaine, any other ingredient of study medication).
2. Pregnancy, breast-feeding or planned pregnancy during the study.
3. Known hypermagnesaemia.
4. Known hypophosphataemia.
5. Clinically significant obstipation, as judged by the investigator.
6. Acute appendicitis.
7. Total intended radiation dose at lips and the anterior oral cavity > 60% of total intended radiation dose at the swallowing process (pharynx, oesophagus).
8. Hyper-fractionated RT.
9. Intended naso-gastral tubes.
10. Primary tumour of the cranial base, brain, oral cavity, lips, naso-pharynx, para-nasal sinuses.
11. Known bone metastases.
12. Reflux oesophagitis 3 months prior to the study.
13. Continuous systemic pain treatment at the beginning of RT. Systemic pain medication for oesophagitis prior to randomisation must not be taken.
14. Concomitant treatment with tetracyclines, cinolone derivatives (ciprofloxacin, ofloxacin, enoxacin, norfloxacin), cheno-desoxycholic acid, sodium fluoride, local anaesthetics (other than those used as study medication).
15. Patients relying on levothyroxine after resection of thyroid carcinoma being hypothyroid and patients relying on levothyroxine due to other reasons not being euthyroid.
16. Artificial nutrition at the beginning of radiation.
17. Drug (licit and illicit) or alcohol abuse which would interfere with the patient's proper completion of the study.
18. Exposure to an investigational product within the last 4 weeks, simultaneous exposure to another investigational product.
19. Lack of ability or willingness to give informed consent.
20. Anticipated non-availability for study visits / procedures.
21. Lack of ability or willingness to keep patient's diary.
22. Lack of willingness to have personal study related data collected, archived or transmitted according to the protocol.
23. Vulnerable subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Time from randomisation to requirement of additional systemic pain medication for oesophagitis (ASPO). | up to 11 weeks

SECONDARY OUTCOMES:
ASPO: WHO analgesic pain ladder | up to 11 weeks
  ASPO = Additional systemic pain medication for oesophagitis
Pain intensity recorded on NRS with scores 0-10 | up to 11 weeks
  NRS = Numeric Rating Scale
Swallowing disorder recorded on NRS with scores 0-10 | up to 11 weeks
  NRS = Numeric Rating Scale
Adapted CTCAE grade | up to 11 weeks
  CTCAE = Common Terminology Criteria for Adverse Events
  Severity of oesophageal symptoms will be evaluated by the investigator according to an adapted CTCAE grading system. In contrast to the original CTCAE classification the adapted version foreseen to be used in this study distinguishes level 2a and 2b.
  2a = symptomatic; altered eating/swallowing; oral supplements indicated; requiring predominantly pureed or soft diet, 2b = symptomatic; altered eating/swallowing; oral supplements indicated; requiring predominantly liquid diet.
Incidence of artificial nutrition due to radiation-induced oesophagitis | up to 11 weeks
Incidence of interruptions of radiation therapy due to radiation-induced oesophagitis | up to 11 weeks
Duration of pain medication intake after the end of Radiation Therapy | up to 11 weeks
Loss of body weight | up to 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Bruns, Dr. med., Principal Investigator — Hannover Medical School; Ursula Petzold, PhD, Study Chair — MEDA Pharma GmbH & Co. KG
Locations (32):
- Austria (2):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Universitätsklinik für Strahlentherapie-Radioonkologie, Innsbruck
- Germany (30):
  - Universitätsklinikum Aachen, Aachen
  - RADIO LOG Strahlentherapie Altötting, Altötting
  - please contact Dr. Ingrid Schwienhorst/MEDA for details, Bad Homburg
  - VIVANTES Klinikum Neukölln, Berlin
  - Strahlenheilkunde Westend, Berlin
  - Franziskus Hospital, Bielefeld
  - Klinik für Hämatologie, Onkologie & Palliativmedizin, Bochum
  - Strahlentherapie Bonn-Rhein-Sieg, Bonn
  - Städtisches Klinikum Braunschweig GmbH, Braunschweig
  - Strahlentherapie Coesfeld, Coesfeld
  - Knappschaftskrankenhaus Dortmund, Dortmund
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - Strahlentherapie - Freising, Freising
  - Kreiskrankenhaus Gummersbach, Gummersbach
  - Universitätsklinikum Halle (Saale), Halle
  - Medizinische Hochschule Hannover, Hanover
  - Kath. Krankenhaus Marienhospital, Herne
  - Universitätsklinikum Leipzig, Leipzig
  - Klinik für Strahlentherapie und Radioonkologie, Marburg
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Gemeinschaftspraxis für Strahlentherapie und Radioonkologie am Klinikum Schwabing, München
  - Klinikum der Universität München, München
  - Paracelsus-Klinik Osnabrück, Osnabrück
  - Paracelsus-Krankenhaus Ruit, Ostfildern
  - Brüderkrankenhaus St. Josef, Paderborn
  - Klinikum Ernst von Bergmann, Potsdam
  - Prosperhospital Recklinghausen, Recklinghausen
  - Universitätsklinikum Rostock AöR, Rostock
  - Klinik für Radioonkologie und Strahlentherapie, Stuttgart